CLINICAL TRIAL: NCT03535649
Title: Clinical Effectiveness and Safety of Vedolizumab Intravenous in Real World Clinical Practice in Ulcerative Colitis Korean Patients: a Multicenter Post-marketing Observational Study
Brief Title: A Study to Assess Clinical Effectiveness and Safety of Vedolizumab Intravenous in Real World Clinical Practice in Ulcerative Colitis (UC) Korean Participants
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5045; U1111-1208-5399 (Other: WHO)
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Colitis, Ulcerative
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vedolizumab: Participants diagnosed with moderate to severe active UC and having failed tumor necrosis factor alpha (TNF alpha) antagonist therapy and who have initiated vedolizumab intravenous treatment between 17 August 2017 and the date when at least 100 cases are collected from approximately 15 participating sites will be observed from the date of UC diagnosis until the date when participant is enrolled into the study or until the end of treatment or death of participants or lost-to-follow up.

SUMMARY:
The purpose of this study is to assess the clinical effectiveness by the clinical response at 6 weeks and the safety of vedolizumab intravenous in UC Korean participants.

DETAILED DESCRIPTION:
This is a post-marketing, non-interventional study of participants with moderate to severe UC. The study will review medical records of participants who have initiated medical treatment with vedolizumab intravenous during the defined eligibility period under routine clinical practice to provide the real world data on the effectiveness and safety of vedolizumab intravenous.

The study will enroll approximately 100 participants. All participants will be enrolled in one observational group: Vedolizumab

Both retrospective and prospective data will be collected in the index period, with prospective data collected for treatment baseline visit and follow up visits.

The multi-center trial will be conducted in Republic of Korea. The overall duration of study will be approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Moderately to severely active UC and having failed TNF-alpha antagonist therapy.

Exclusion Criteria:

1. Was treated with vedolizumab intravenous outside of the locally approved label in South Korea.
2. Was enrolled in an Interventional Intestinal Bowel Disease clinical trial at time of using vedolizumab intravenous.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with moderate to severe UC, having failed TNF-alpha antagonist therapy and who have initiated treatment with vedolizumab intravenous between 17 August 2017 and up until 100 participants are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (15):
- South Korea (15):
  - Dankook University Hospital, Cheonan-si, Chungcheongnam-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Inje University Haeundae Paik Hospita, Busan
  - Kyungpook National University Hospital, Daegu
  - Youngnam University Hospital, Daegu
  - Goo Hospital, Daegu
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in South Korea from 17 August 2017 to 18 December 2018.
Pre-assignment Details: Participants with a diagnosis of moderately to severely active ulcerative colitis (UC), having failed tumor necrosis factor-alpha (TNF-alpha) antagonist therapy and who have been prescribed vedolizumab intravenously under standard clinical practice were enrolled in this observational study.
Groups:
- Vedolizumab: Participants diagnosed with moderate to severe active UC, having failed TNF-alpha antagonist therapy and received vedolizumab intravenous treatment were observed under standard clinical practice until the end of treatment or death of participants or lost to-follow up, whichever occurred first.
Period: Overall Study
Arm/Group | Vedolizumab
Started | 105
Completed | 105
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) consisted all enrolled participants who received at least one documented dose of study medication.
Arm/Group | Vedolizumab
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Korea, Republic Of | 105
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: Number analyzed signifies participants for whom body weight data was available at baseline.
  kilogram (kg)
    number analyzed (Participants) | 90
    (all) | 61.4 (12.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Population: Number analyzed signifies participants for whom BMI was available at baseline.
  kilogram per square meter (kg/m^2)
    number analyzed (Participants) | 88
    (all) | 22.0 (3.47)
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 4
  Former smoker | 31
  Never smoked | 62
  Unknown | 8
Family History [Count of Participants; unit: Participants]
  Crohn's disease | 0
  UC- Siblings | 2
  UC- Parent | 1
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 5
  Diabetes mellitus | 2
  Autoimmune hepatitis | 1
  Rheumatoid arthritis | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response at Week 6 Based on Partial Mayo Score
Description: Clinical response based on partial Mayo score was defined as a reduction of at least 3 points and a decrease of at least 30 percent (%) from the baseline Mayo score, with a decrease of at least 1 point on the rectal bleeding subscale, or an absolute rectal bleeding score of 0 or 1. Mayo score was an instrument designed to measure disease activity of UC. Partial Mayo score consisted of 3 sub-scores: stool frequency, most severe rectal bleeding of the day, and global assessment by physician, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed to give a total score range of 0 to 9; where higher score indicated more severe disease.
Time Frame: Week 6
Population: The full analysis set (FAS) consisted all enrolled participants who received at least one dose of study medication and had active disease at baseline. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab
Number analyzed (Participants) | 77
percentage of participants | 55.8

2. Primary Outcome: Percentage of Participants With Adverse Events of Special Interests (AESIs) and Serious Adverse Events (SAEs)
Time Frame: From the index date (date when vedolizumab treatment was initiated) until the end of treatment, lost to follow-up or death (up to 15 months)
Population: The SAS consisted all enrolled participants who received at least one documented dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab
Number analyzed (Participants) | 105
percentage of participants
  AESIs | 4.76
  SAEs | 4.76

3. Primary Outcome: Percentage of Participants With Pregnancy During the Study
Time Frame: as for outcome 2
Population: The SAS consisted all enrolled participants who received at least one documented dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab
Number analyzed (Participants) | 105
percentage of participants | 0.00

4. Secondary Outcome: Percentage of Participants With Clinical Response at Week 14 Based on Partial Mayo Score
Description: Clinical response was defined as a reduction of at least 3 points and a decrease of at least 30% from the baseline mayo score, with a decrease of at least 1 point on the rectal bleeding subscale, or an absolute rectal bleeding score of 0 or 1. Mayo score was an instrument designed to measure disease activity of UC. Partial Mayo score consisted of 3 sub-scores: stool frequency, most severe rectal bleeding of the day, endoscopic findings and global assessment by physician, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher scores indicated more severe disease.
Time Frame: Week 14
Population: The FAS consisted all enrolled participants who received at least one dose of study medication and had active disease at baseline. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab
Number analyzed (Participants) | 71
percentage of participants | 73.2

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 6 and Week 14 Based on Partial Mayo Score
Description: Clinical remission was defined as a total mayo score of less than or equal to (<=) 2 with no sub-score greater than (>) 1. Mayo score was an instrument designed to measure disease activity of UC. Partial Mayo score consisted of 3 sub-scores: stool frequency, most severe rectal bleeding of the day, and global assessment by physician, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed to give a total score range of 0 to 9; where higher score indicated more severe disease.
Time Frame: Weeks 6 and 14
Population: The FAS consisted all enrolled participants who received at least one dose of study medication and had active disease at baseline. Here, n (number analyzed) signifies number of participants who were analyzed at specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab
Number analyzed (Participants) | 77
percentage of participants
  Week 6 | 18.2
  Week 14: number analyzed (Participants) | 71
  Week 14 | 39.4

6. Secondary Outcome: Percentage of Participants With Mucosal Healing at Weeks 6 and 14
Description: Mucosal healing was defined as Mayo endoscopic sub-score of 0 or 1 compared to baseline. Mayo score was an instrument designed to measure disease activity of UC. Endoscopic findings was a sub-score of complete Mayo score, which ranges from 0 to 3 (0= Normal or inactive disease; 1= Mild disease; 2= Moderate disease; 3= Severe disease), with higher scores indicating more severe disease.
Time Frame: Weeks 6 and 14
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab
Number analyzed (Participants) | 59
percentage of participants
  Week 6: number analyzed (Participants) | 9
  Week 6 | 22.2
  Week 14 | 49.2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are adverse events that started after the first dose of study drug (index date) until end of treatment, lost to follow-up or death (up to 15 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vedolizumab
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 5/105
Other Adverse Events (participants affected / at risk) | 16/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vedolizumab (N=105)
Colitis ulcerative (Gastrointestinal disorders) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Adenoiditis (Infections and infestations) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vedolizumab (N=105)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2)
Colitis ulcerative (Gastrointestinal disorders) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Cytomegalovirus syndrome (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT03535649/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT03535649/SAP_001.pdf